CLINICAL TRIAL: NCT01230749
Title: A Double-Blind, Randomized, Placebo- and Active Comparator-Controlled, 4-Week Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Oral Doses of JNJ-41443532 in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study of Multiple Oral Doses of JNJ-41443532 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017401; 41443532EDI2001 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2010-10-22; First posted 2010-10-29 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Diabetes Mellitus; Hyperglycemia; JNJ-41443532; Pioglitazone; Placebo
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hyperglycemia | interventions — JNJ-41443532; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- JNJ-41443532 250 mg (Experimental): Participants will receive JNJ-41443532 250 mg in morning and evening for 28 days.
  Interventions: Drug: JNJ-41443532; Drug: Placebo
- JNJ-41443532 1000 mg (Experimental): Participants will receive JNJ-41443532 1000 mg (4 X 250 mg) in morning and evening for 28 days.
  Interventions: Drug: JNJ-41443532; Drug: Placebo
- Pioglitazone (Active Comparator): Participants will receive pioglitazone 30 mg in morning for 28 days.
  Interventions: Drug: Pioglitazone 30 mg; Drug: Placebo
- Placebo (Placebo Comparator): Participants will receive matching placebo for JNJ-41443532 and pioglitazone for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-41443532 — Participants will receive JNJ-41443532 tablet(s) orally in JNJ-41443532 250 mg arm (1 X 250 mg) and JNJ-41443532 1000 mg arm (4 X 250 mg) in morning and evening, for 28 days.
  Arms: JNJ-41443532 1000 mg; JNJ-41443532 250 mg
Drug: Pioglitazone 30 mg — Participants will receive tablet pioglitazone 30 mg orally in morning for 28 days.
  Arms: Pioglitazone
Drug: Placebo — Participants will receive matching placebo tablets of JNJ-41443532 and/or matching placebo tablets of pioglitazone orally as per the assigned arms.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (what the body does to the medication) and pharmacodynamics (what the medication does to the body) of treatment with JNJ-41443532 relative to treatment with placebo in type 2 diabetes mellitus participants.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), double-blind (neither investigator nor participant knows the treatment that the participant receives), multicenter (study conducted at multiple sites), and placebo (an inactive substance that is compared with a medication to test whether the medication has a real effect in a clinical study) and active comparator (an established effective treatment that is compared with a medication to test whether the medication has a real effect in a clinical study) controlled study (placebo or active comparator is compared with the study medication to test whether the study medication has a real effect in clinical study). The study consists of 4 phases: screening phase (45 days before administration of study medication); pre-dosing run-in phase (a phase before a clinical study is commenced when no treatment is given. In this study, participant's glucose level will be observed during run-in-phase: days 15 to 1 before administration of study medication); treatment phase, and follow-up phase (7 to 10 days after the last dose of the study medication). Approximately 88 participants will be enrolled in this study. All participants will be randomly assigned to 4 treatment arms: JNJ-41443532 250 mg; JNJ-41443532 1000 mg; pioglitazone arm; and placebo. Safety evaluations will include assessment of adverse events including ocular assessments, clinical laboratory tests, electrocardiogram, vital signs, and physical examination which will be monitored throughout the study. The maximum study duration for each participant will be approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Type 2 Diabetes Mellitus (T2DM) for at least 3 months prior screening
* On a stable treatment regimen for at least 2 months prior screening
* Medically stable on the basis of physical examination, medical history, and clinical laboratory tests performed at screening and 2 days before administration of the study medication
* Fasting plasma glucose (FPG) concentrations between 140 mg/dL and 270 mg/dL on 2 days before administration of the study medication
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

* History of other types of diabetes and complications or secondary forms of diabetes
* History of eating disorder or recent significant changes in body weight (ie, more or equal to 5 percent over 3 months prior to screening) due to dieting or nutritional treatments
* Taking antihyperglycemic agents (insulin, exenatide, and liraglutide) within 6 months or thiazolidinedione within 3 months of 2 days before administration of the study medication
* Clinically significant abnormal electrocardiogram
* History of, or currently active, significant illness or medical disorders, retinal disease, tuberculosis
* Clinically important serious infection, positive for serology at screening (hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus antibodies)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 89 participants were enrolled at 7 study sites in United States.
Pre-assignment Details: 89 participants were randomly assigned to 4 treatment groups (Placebo: 22; Pioglitazone 30 mg: 22; JNJ41443532 250 mg: 23, and JNJ41443532 1000 mg: 22) and all participants received at least one dose of the study medication.
Groups:
- Placebo: Participants received placebo tablets orally, twice a day for 29 days.
- Pioglitazone 30 mg: Participants received pioglitazone 30 mg tablet orally, once a day for 29 days.
- JNJ41443532 250 mg: Participants received JNJ-41443532 250 mg tablet orally, twice a day for 29 days.
- JNJ41443532 1000 mg: Participants received JNJ-41443532 1000 mg (4 X 250 mg tablet) orally, twice a day for 29 days.
Period: Overall Study
Arm/Group | Placebo | Pioglitazone 30 mg | JNJ41443532 250 mg | JNJ41443532 1000 mg
Started | 22 | 22 | 23 | 22
Completed | 22 | 20 | 21 | 20
Not Completed | 0 | 2 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Fasting glucose more than 270 mg/dL | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pioglitazone 30 mg | JNJ41443532 250 mg | JNJ41443532 1000 mg | Total
Number analyzed (Participants) | 22 | 22 | 23 | 22 | 89
Age Continuous [Mean (Standard Deviation); unit: years] | 52.7 (8.93) | 54.5 (8.93) | 51.7 (7.06) | 57.1 (6.03) | 54 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 7 | 11 | 34
  Male | 13 | 15 | 16 | 11 | 55

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Day -1) to Day 28 in Twenty-Four-Hour Weighted Average Glucose (24-Hour WAG)
Description: Difference is calculated as the change in 24-hour WAG in Least Square Mean (LSM) from baseline to Day 28 of each treatment group (pioglitazone, JNJ-41443532 250 mg, JNJ-41443532 1000 mg, and placebo). The statistical analyses shows the treatment differences (ie, each study medication group minus placebo) in the LSM change. 24-hour WAG is defined as the area under the plasma glucose concentration time curve over 0 to 24 hours, divided by 24.
Time Frame: From baseline (Day -1) to Day 28
Population: Analyses included all participants who received at least 1 dose of JNJ-41443532 or placebo and had at least 1 pharmacodynamic assessment posttreatment.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- Placebo: Participants received placebo orally, twice a day for 29 days
Arm/Group | Pioglitazone 30 mg | JNJ41443532 250 mg | JNJ41443532 1000 mg | Placebo
Number analyzed (Participants) | 20 | 21 | 20 | 22
mg/dL | -18.88 (7.74) [-46.792 to -8.008] | -11.95 (7.33) [-39.801 to -1.142] | -4.72 (7.56) [-32.635 to 6.151] | 8.52 (7.23)
Statistical Analysis 1: Comparison: Pioglitazone 30 mg vs Placebo; Test type: Superiority or Other; p = 0.006, ANCOVA; Difference in LSM = -27.40, 95% CI 2-sided [-46.792 to -8.008]
Statistical Analysis 2: Comparison: JNJ41443532 250 mg vs Placebo; Test type: Superiority or Other; p = 0.038, ANCOVA; Difference in LSM = -20.47, 95% CI 2-sided [-39.801 to -1.142]
Statistical Analysis 3: Comparison: JNJ41443532 1000 mg vs Placebo; Test type: Superiority or Other; p = 0.178, ANCOVA; Difference in LSM = -13.24, 95% CI 2-sided [-32.635 to 6.151]

2. Secondary Outcome: Change From Baseline to Day 28 in Fasting Plasma Glucose (FPG)
Description: Difference is calculated as the change in FPG in Least Square Mean (LSM) from baseline to Day 28 of each treatment group (pioglitazone, JNJ-41443532 250 mg, JNJ-41443532 1000 mg, and placebo). The statistical analyses shows the treatment differences (ie, each study medication group minus placebo) in the LSM change.
Time Frame: From baseline to Day 28
Population: Analyses included all participants who received at least 1 dose of JNJ-41443532 or placebo and had at least 1 pharmacodynamic assessment posttreatment. Two participants (1 in JNJ-41443532 250-mg group and 1 in Pioglitazone group) were excluded from the analysis because a blood sample for FPG was not collected on Day 28.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone 30 mg | JNJ41443532 250 mg | JNJ41443532 1000 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
mg/dL | -14.57 (7.93) [-47.606 to -8.957] | -8.26 (7.47) [-41.154 to -2.786] | -4.00 (7.29) [-36.860 to 1.431] | 13.71 (7.23)
Statistical Analysis 1: Comparison: Pioglitazone 30 mg vs Placebo; Test type: Superiority or Other; p = 0.005, ANCOVA; Difference in LSM = -28.28, 95% CI 2-sided [-47.606 to -8.957]
Statistical Analysis 2: Comparison: JNJ41443532 250 mg vs Placebo; Test type: Superiority or Other; p = 0.025, ANCOVA; Difference in LSM = -21.97, 95% CI 2-sided [-41.154 to -2.786]
Statistical Analysis 3: Comparison: JNJ41443532 1000 mg vs Placebo; Test type: Superiority or Other; p = 0.069, ANCOVA; Difference in LSM = -17.71, 95% CI 2-sided [-36.860 to 1.431]

3. Secondary Outcome: Change From Baseline to Day 28 in Insulin Secretion
Description: Difference is calculated as the change in insulin secretion in Least Square Mean (LSM) from baseline to Day 28 of each treatment group (pioglitazone, JNJ-41443532 250 mg, JNJ-41443532 1000 mg, and placebo). The statistical analyses shows the treatment differences (ie, each study medication group minus placebo) in the LSM change. Insulin secretion is measured by the absolute change in Homeostasis Model Assessment of steady state islet beta cell (HOMA-%B). HOMA-%B calculated as: (360 multiplied by Insulin [pmol/L]) divided by ([Glucose {mg/dL} minus 63] multiplied by 6.945). Higher value is better (signifies improvement relative to baseline).
Time Frame: From baseline to Day 28
Population: Analyses included all participants who received at least 1 dose of JNJ-41443532 or placebo and had at least 1 pharmacodynamic assessment posttreatment. Two participants (1 in JNJ-41443532 250-mg group and 1 in Pioglitazone group) were excluded from the analysis because a blood sample for HOMA-%B was not collected on Day 28.
Measure: Least Squares Mean (Standard Error); unit: HOMA-B score
Arm/Group | Pioglitazone 30 mg | JNJ41443532 250 mg | JNJ41443532 1000 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
HOMA-B score | -4.00 (4.644) [-15.852 to 26.334] | 6.94 (4.415) [3.146 to 45.370] | -0.89 (4.301) [-8.022 to 34.107] | -6.76 (4.255)
Statistical Analysis 1: Comparison: Pioglitazone 30 mg vs Placebo; Test type: Superiority or Other; p = 0.628, ANCOVA; Difference in LSM = 2.76, 95% CI 2-sided [-8.542 to 14.054]
Statistical Analysis 2: Comparison: JNJ41443532 250 mg vs Placebo; Test type: Superiority or Other; p = 0.018, ANCOVA; Difference in LSM = 13.70, 95% CI 2-sided [2.392 to 25.008]
Statistical Analysis 3: Comparison: JNJ41443532 1000 mg vs Placebo; Test type: Superiority or Other; p = 0.303, ANCOVA; Difference in LSM = 5.87, 95% CI 2-sided [-5.417 to 17.148]

4. Secondary Outcome: Change From Baseline to Day 28 in Insulin Resistance
Description: Difference is calculated as the change in insulin resistance in Least Square Mean (LSM) from baseline to Day 28 of each treatment group (pioglitazone, JNJ-41443532 250 mg, JNJ-41443532 1000 mg, and placebo). The statistical analyses shows the treatment differences (ie, each study medication group minus placebo) in the LSM change. Insuline sensitivity is measured by absolute change in Homeostasis Model Assessment of insulin resistance (HOMA-IR). Insulin sensitivity is HOMA-%S and HOMA-IR is the reciprocal of HOMA-%S. HOMA-IR calculated as: (Glucose [mg/dL]) multiplied by Insulin [pmol/L]) divided by (405 multiplied by 6.945). Lower value is better (signifies improvement relative to baseline).
Time Frame: From baseline to Day 28
Population: Analyses included all participants who received at least 1 dose of JNJ-41443532 or placebo and had at least 1 pharmacodynamic assessment posttreatment. Two participants (1 in JNJ-41443532 250-mg group and 1 in Pioglitazone group) were excluded from the analysis because a blood sample for HOMA-IR was not collected on Day 28.
Measure: Least Squares Mean (Standard Error); unit: HOMA-IR score
Arm/Group | Pioglitazone 30 mg | JNJ41443532 250 mg | JNJ41443532 1000 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 20 | 21
HOMA-IR score | -1.52 (0.739) [-48.370 to -7.180] | 0.07 (0.689) [-24.534 to 16.542] | -0.35 (0.675) [-30.592 to 10.615] | 0.33 (0.666)
Statistical Analysis 1: Comparison: Pioglitazone 30 mg vs Placebo; Test type: Superiority or Other; p = 0.041, ANCOVA; Difference in LSM = -1.86, 95% CI 2-sided [-3.634 to -0.082]
Statistical Analysis 2: Comparison: JNJ41443532 250 mg vs Placebo; Test type: Superiority or Other; p = 0.769, ANCOVA; Difference in LSM = -0.26, 95% CI 2-sided [-2.033 to 1.509]
Statistical Analysis 3: Comparison: JNJ41443532 1000 mg vs Placebo; Test type: Superiority or Other; p = 0.444, ANCOVA; Difference in LSM = -0.69, 95% CI 2-sided [-2.463 to 1.091]

5. Secondary Outcome: Change From Baseline to Day 28 in Systemic Levels of Interleukin 6 (IL-6)
Description: Difference is calculated as the geometric mean change in IL-6 from baseline to Day 28 of each treatment group (JNJ-41443532 250 mg, JNJ-41443532 1000 mg, and placebo). The statistical analyses shows the treatment differences (ie, each study medication group minus placebo) in the geometric mean change. IL-6 is a systemic inflammatory markers and is an independent predictors of insulin resistance and progression to type 2 diabetes mellitus. IL-6 was not measured for pioglitazone guoup. The unit of IL-6 is picograms per milliliter (pg/mL).
Time Frame: From baseline to Day 28
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: pg/mL
Arm/Group | JNJ41443532 250 mg | JNJ41443532 1000 mg | Placebo
Number analyzed (Participants) | 21 | 20 | 22
pg/mL | 0.86 (0.85) [71.031 to 127.324] | 0.81 (0.34) [66.567 to 121.403] | 0.91 (0.71)
Statistical Analysis 1: Comparison: JNJ41443532 250 mg vs Placebo; Test type: Superiority or Other; p = 0.774, ANCOVA; GMR mulitplied by 100 percent = 95.10, 90% CI 2-sided [71.031 to 127.324]
Statistical Analysis 2: Comparison: JNJ41443532 1000 mg vs Placebo; Test type: Superiority or Other; p = 0.555, ANCOVA; GMR multiplied by 100 percent = 89.90, 90% CI 2-sided [66.567 to 121.403]

6. Secondary Outcome: Change From Baseline to Day 28 in Systemic Levels of Interleukin 18 (IL-18)
Description: Difference is calculated as the geometric mean change in IL-18 from baseline to Day 28 of each treatment group (JNJ-41443532 250 mg, JNJ-41443532 1000 mg, and placebo). The statistical analyses shows the treatment differences (ie, each study medication group minus placebo) in the geometric mean change. IL-18 was not measured for pioglitazone group. The unit of IL-18 is picograms per milliliter (pg/mL)
Time Frame: From baseline to Day 28
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: pg/mL
Arm/Group | JNJ41443532 250 mg | JNJ41443532 1000 mg | Placebo
Number analyzed (Participants) | 21 | 20 | 22
pg/mL | 1.02 (0.16) [93.217 to 107.647] | 1.03 (0.12) [94.179 to 108.700] | 1.02 (0.15)
Statistical Analysis 1: Comparison: JNJ41443532 250 mg vs Placebo; Test type: Superiority or Other; p = 0.968, ANCOVA; GMR multiplied by 100 percent = 100.17, 90% CI 2-sided [93.217 to 107.647]
Statistical Analysis 2: Comparison: JNJ41443532 1000 mg vs Placebo; Test type: Superiority or Other; p = 0.785, ANCOVA; GMR multiplied by 100 percent = 101.18, 90% CI 2-sided [94.179 to 108.700]

7. Secondary Outcome: Change From Baseline to Day 28 in Systemic Levels of C-Reactive Protein (CRP)
Description: Difference is calculated as the geometric mean change in CRP from baseline to Day 28 of each treatment group (JNJ-41443532 250 mg, JNJ-41443532 1000 mg, and placebo). The statistical analyses shows the treatment differences (ie, each study medication group minus placebo) in the geometric mean change. CRP was not measured for pioglitazone group.
Time Frame: From baseline to Day 28
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: mg/dL
Arm/Group | JNJ41443532 250 mg | JNJ41443532 1000 mg | Placebo
Number analyzed (Participants) | 21 | 20 | 22
mg/dL | 1.12 (0.56) [100.275 to 177.115] | 0.86 (0.30) [76.260 to 135.942] | 0.84 (0.63)
Statistical Analysis 1: Comparison: JNJ41443532 250 mg vs Placebo; Test type: Superiority or Other; p = 0.097, ANCOVA; GMR multiplied by 100 percent = 133.27, 90% CI 2-sided [100.275 to 177.115]
Statistical Analysis 2: Comparison: JNJ41443532 1000 mg vs Placebo; Test type: Superiority or Other; p = 0.917, ANCOVA; GMR mulitplied by 100 percent = 101.82, 90% CI 2-sided [76.260 to 135.942]

8. Secondary Outcome: Change From Baseline to Day 29 in Body Weight
Description: Difference is calculated as the change in body weight in Least Square Mean (LSM) from baseline to Day 29 of each treatment group (pioglitazone, JNJ-41443532 250 mg, JNJ-41443532 1000 mg, and placebo). The statistical analyses shows the treatment differences (ie, each study medication group minus placebo) in the LSM change.
Time Frame: From baseline to Day 29
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Pioglitazone 30 mg | JNJ41443532 250 mg | JNJ41443532 1000 mg | Placebo
Number analyzed (Participants) | 20 | 21 | 20 | 22
Kilograms | -0.75 (0.35) [-0.408 to 1.323] | -1.18 (0.34) [-0.838 to 0.904] | -0.19 (0.34) [0.150 to 1.892] | -1.21 (0.32)
Statistical Analysis 1: Comparison: Pioglitazone 30 mg vs Placebo; Test type: Superiority or Other; p = 0.295, ANCOVA; Difference in LSM = 0.46, 95% CI 2-sided [-0.408 to 1.323]
Statistical Analysis 2: Comparison: JNJ41443532 250 mg vs Placebo; Test type: Superiority or Other; p = 0.941, ANCOVA; Difference in LSM = 0.03, 95% CI 2-sided [-0.838 to 0.904]
Statistical Analysis 3: Comparison: JNJ41443532 1000 mg vs Placebo; Test type: Superiority or Other; p = 0.022, ANCOVA; Difference in LSM = 1.02, 95% CI 2-sided [0.150 to 1.892]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | Pioglitazone 30 mg | JNJ41443532 250 mg | JNJ41443532 1000 mg
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/23 | 1/22
Other Adverse Events (participants affected / at risk) | 6/22 | 7/22 | 9/23 | 4/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | Pioglitazone 30 mg (N=22) | JNJ41443532 250 mg (N=23) | JNJ41443532 1000 mg (N=22)
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | Pioglitazone 30 mg (N=22) | JNJ41443532 250 mg (N=23) | JNJ41443532 1000 mg (N=22)
Vision Blurred (Eye disorders) | 2 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Dry Mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 2 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 4 | 2 | 4 | 1
Paraesthesia (Nervous system disorders) | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 2 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days